CLINICAL TRIAL: NCT07363707
Title: A Comparative Study of the Effect of Dapagliflozin Versus Empagliflozin ,Added to Metformin, on NAFLD in Patients With Type 2 Diabetes
Brief Title: A Study Between Dapagliflozin and Empagliflozin Effect on NAFLD in Patients With Type 2 Diabetes.
Acronym: (Dapa)& (Empa)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Beni-Suef University (Other)
Responsible Party: Principal Investigator, Aya Allah Emad ELdin Abdelazeem Abdelmotaleb, bachelor of clinical pharmacy, Beni-Suef University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: effect of Dapa &Empa on NAFLD
Record Dates: First submitted 2025-12-19; First posted 2026-01-23 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2025-12

CONDITIONS: NAFLD (Nonalcoholic Fatty Liver Disease)
Keywords: Dapagliflozin and Empagliflozin
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — dapagliflozin; Metformin

STUDY DESIGN:
Intervention Model Description: In this prospective randomized controlled trial, a number of 108 patients of MASLD and T2DM were enrolled into 2 equal groups to either receive Dapa 10mg /day(control group; n=54) or or Empa 25mg/day (n = 54), in addition to conventional therapy (metformin) for 6 months.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dapagliflozin (Active Comparator)
  Interventions: Drug: Dapagliflozin + Metformin
- Empagliflozin (Active Comparator)
  Interventions: Drug: Empa

INTERVENTIONS:
Drug: Dapagliflozin + Metformin — name and concentration of drug ( Dapagliflozin 10 mg)
  Arms: Dapagliflozin
Drug: Empa — name and concentration of drug Empagliflozin 25
  Arms: Empagliflozin

SUMMARY:
The goal of this clinical trial is to learn if drugs Dapagliflozin and Empagliflozin work to treat NAFLD in Type 2 diabetes patients. It will also learn about the safety of drugs dapagliflozin and empagliflozin. The main questions it aims to answer are:

Do drug dapagliflozin and empagliflozin lower the NAFLD degree for participants? What medical problems do participants have when taking the drugs dapagliflozin and empagliflozin?

Researchers will compare drug dapagliflozin to empagliflozin to see which of them more effective to treat NAFLD.

Participants will:

Take drug dapagliflozin or empaglifloin every day for 6 months Visit the clinic once every 2 weeks for checkups and tests Keep a diary of their symptoms and the number of times they use a rescue inhaler

DETAILED DESCRIPTION:
Type 2 Diabetes Mellitus (T2DM) and Metabolic Dysfunction-Associated Steatotic Liver Disease (MASLD) are two chronic, interconnected metabolic disorders that affect millions of individuals worldwide. MASLD is currently the most prevalent chronic liver disease, with a global burden of 17 % to 46% of chronic liver disease cases. Patients with DM2 have a very high prevalence of MASLD, which can vary from 40% to 60%. In clinical settings, MASLD has been reported to share similar pathophysiological mechanisms (such as insulin resistance, defective hepatic lipid profile, and abnormal triglyceride metabolism) with type 2 diabetes and is strongly associated with it . It has been revealed that MASLD increases the risk of type 2 diabetes incidents by approximately twofold. Therefore, reducing the prevalence of MASLD could help mitigate the impact of type 2 diabetes to some extent. SGLT2 inhibitors are promising for MASLD and T2DM because they improve glucose control, promote weight loss, and have direct beneficial effects on the liver, such as reducing liver fat and inflammation. So, Sodium-Glucose Transport Protein 2 (SGLT-2) inhibitors would be promising therapeutic agents for treatment of MASLD/ Nonalcoholic Steatohepatitis (NASH) patients. Therefore, great interest should be provided towards SGLT-2i treatment that contributes to alleviation of MASLD by reduction of hyperglycaemia, improvement of systematic insulin resistance, elevation of caloric loss and reduction of body weight mostly due to glycosuria.

The management of (T2DM) and (MASLD) involves a multifaceted approach that targets the underlying pathophysiology of both diseases. Management strategies typically focus on controlling blood glucose levels, improving insulin sensitivity, and addressing the hepatic fat accumulation and inflammation that characterize MASLD.(12) Nevertheless, animal and human studies on incretin mimetics, glucagon-like peptide-1 receptor agonists (GLP-1 RA) approved for T2DM treatment, have provided indirect evidence that they may also ameliorate progression of MASLD/NASH, over other antidiabetic types in T2DM patients with MASLD. Therefore, newer antidiabetic agents with an additive MASLD-lowering effect would be of great interest.

Sodium-glucose co-transporter 2 (SGLT-2) inhibitors are a promising oral treatment for T2D either as monotherapy or in combination with other antidiabetic agents. In addition to their anti-hyperglycemic effects and ability to reduce body weight, SGLT-2i seem to exert potent antioxidant and anti-inflammatory effects, making them promising candidates for MASLD treatment. SGLT2 inhibitors induce a series of modifications that have the potential to improve the liver condition in individuals with MASLD; they improve glycemic profile, reduce visceral adipose tissue, increase plasma adiponectin levels, and decrease uric acid levels; they also diminish oxidative stress and systemic inflammation and increase glucacon levels. Short and long-term follow-up studies should elucidate the role of these drugs in the prevention and attenuation of MASLD progression in early stages. The main aim of the present study is to compare the effects of two (SGLT-2)i , Dapa versus Empa, added to metformin) on liver steatosis and fibrosis for 6 monthsin patients with MASLD and T2D .

ELIGIBILITY:
Inclusion Criteria:

* Adults from 18 years old, male or female type 2 diabetic NAFLD patients.

Exclusion Criteria:

* People who have chronic liver disease,
* Hepatitis C virus (HCV) patients or those treated for HCV,
* History of autoimmune disease,
* Drugs that cause steatohepatitis
* and alcoholic patients will be excluded.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2023-08-27 (Actual); Study Completion 2024-03-01 (Actual)

PRIMARY OUTCOMES:
Fibro scan, as well as the changes in FIB4 score and Full lipid profile (total cholesterol, LDL, HDL, VLDL, and triglyceride). | at zero month and after 6 six months
  by using Fibro scan(Controlled Attenuation Parameter (CAP) The liver CAP score assesses fatty change (S1, S2, S3 grades), and Elasticity Score (E) kilopascals (kPa)) as well as the changes in FIB4 score (has no units; it's a calculated index (a number) derived from blood tests (AST, ALT, platelets) and age) and Full lipid profile (total cholesterol, LDL, HDL, VLDL and triglyceride (mg/dL) ) from baseline to six months in the two groups.
  In a lipid profile, mg/dL stands for milligrams per deciliter. This is the standard unit of measurement used to express the concentration of cholesterol and fats in the blood.
  What it Measures
  The measurement indicates how many milligrams (mg) of a specific lipid are found in one deciliter (dL) of blood. A lipid profile typically reports several components using this unit:
  Total Cholesterol: The overall amount of cholesterol (mg) in your blood(dl). LDL (Low-Density Lipoprotein) HDL (High-Density Lipoprotein) VLDLvery Low-Density Lipopr Triglycerides

CONTACTS AND LOCATIONS:
Locations (1):
- Beni Suef University Hospital, Cairo, Egypt

REFERENCES:
- [Background] 11. Androutsakos T, Nasiri-Ansari N, Bakasis A-D, Kyrou I, Efstathopoulos E, Randeva HS, et al. SGLT-2 inhibitors in NAFLD: expanding their role beyond diabetes and cardioprotection. International journal of molecular sciences. 2022;23(6):3107. 12. Abdel-Rahman RF. Non-alcoholic fatty liver disease: epidemiology, pathophysiology and an update on the therapeutic approaches. Asian Pacific Journal of Tropical Biomedicine. 2022;12(3):99-114. 13. Athyros VG, Polyzos SA, Kountouras J, Katsiki N, Anagnostis P, Doumas M, et al. Non-Alcoholic Fatty Liver Disease Treatment in Patients with Type 2 Diabetes Mellitus; New Kids on the Block. Current vascular pharmacology. 2020;18(2):172-81. 14. Mohsen M, Elberry AA, Mohamed Rabea A, Abdelrahim ME, Hussein RR. Saxagliptin and vildagliptin lowered albuminuria in patients with diabetes and hypertension independent on glycaemic control. International Journal of Clinical Practice. 2021;75(3):e13769. 15. Xia C, Goud A, D'Souza J, Dahagam C, Rao X, Rajagopalan S, et al. DPP4 inhibitors and cardiovascular outcomes: safety on heart failure. Heart failure reviews. 2017;22:299-304. 16. Niezen S, Diaz del Castillo H, Mendez Castaner LA, Fornoni A. Safety and efficacy of antihyperglycaemic agents in diabetic kidney disease. Endocrinology, diabetes & metabolism. 2019;2(3):e00072. 17. Scheen A. Beneficial effects of SGLT2 inhibitors on fatty liver in type 2 diabetes: a common comorbidity associated with severe complications. Diabetes & metabolism. 2019;45(3):213-23. 18. Ciardullo S, Vergani M, Perseghin G. Nonalcoholic Fatty Liver Disease in Patients with Type 2 Diabetes: Screening, Diagnosis, and Treatment. Journal of Clinical Medicine. 2023;12(17):5597.
- [Background] 1. Bica C, Sandu C, Suceveanu AI, Sarbu E, Stoica RA, Gherghiceanu F, et al. Non-alcoholic fatty liver disease: A major challenge in type 2 diabetes mellitus. Experimental and Therapeutic Medicine. 2020;20(3):2387-91. 2. Das C, Tripathy D, Swain S, Sudhakaran N, Uthansingh K, Mallick P, et al. Effect of Dapa on type 2 diabetes mellitus with nonalcoholic fatty liver disease: a single-center survey. Cureus. 2021;13(5). 3. Almahmoud MH, Al Khawaja NM, Alkinani A, Khader Y, Ajlouni KM. Prevalence of fatty liver disease and its associated factors among Jordanian patients with type 2 diabetes mellitus: A cross-sectional study. Annals of Medicine and Surgery. 2021;68:102677. 4. Tanase DM, Gosav EM, Costea CF, Ciocoiu M, Lacatusu CM, Maranduca MA, et al. The intricate relationship between type 2 diabetes mellitus (T2DM), insulin resistance (IR), and nonalcoholic fatty liver disease (NAFLD). Journal of diabetes research. 2020;2020(1):3920196. 5. Targher G, Corey KE, Byrne CD, Roden M. The complex link between NAFLD and type 2 diabetes mellitus-mechanisms and treatments. Nature reviews Gastroenterology & hepatology. 2021;18(9):599-612. 6. Stefan N, Cusi K. A global view of the interplay between non-alcoholic fatty liver disease and diabetes. The lancet Diabetes & endocrinology. 2022;10(4):284-96. 7. Younossi ZM. Non-alcoholic fatty liver disease-a global public health perspective. Journal of hepatology. 2019;70(3):531-44. 8. Loomba R, Abraham M, Unalp A, Wilson L, Lavine J, Doo E, et al. Association between diabetes, family history of diabetes, and risk of nonalcoholic steatohepatitis and fibrosis. Hepatology. 2012;56(3):943-51. 9. Musso G, Gambino R, Cassader M, Pagano G. Meta-analysis: natural history of non-alcoholic fatty liver disease (NAFLD) and diagnostic accuracy of non-invasive tests for liver disease severity. Annals of medicine. 2011;43(8):617-49. 10. Popoviciu MS, Păduraru L, Rahman MM, Supti FA, Stoica RA, Reurean-Pintilei D, et al. The effects of SGLT2 inhibitor